CLINICAL TRIAL: NCT00307554
Title: Assess Lot-to-lot Consistency of 3 Lots (Double Blind Design) of GlaxoSmithKline Biologicals' 10-valent Pneumococcal Vaccine and Evaluate Non-inferiority to Prevenar™ (Single Blind Design) When Administered as 3-dose Primary Immunization Course Before 6 Months of Age
Brief Title: A Lot-to-lot Consistency (3 Lots of GSK Biologicals' 10-valent Pneumococcal Conjugate Vaccine) & Non-inferiority Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 105553
Record Dates: First submitted 2006-03-08; First posted 2006-03-28 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Streptococcal
MeSH Terms: conditions — Streptococcal Infections | interventions — Pneumococcal Vaccines

INTERVENTIONS:
Biological: Pneumococcal (vaccine)

SUMMARY:
Evaluate lot-to-lot consistency, safety and reactogenicity of 3 doses of GSK Biologicals' 10-valent pneumococcal conjugate vaccine and non-inferiority with respect to Prevenar.

DETAILED DESCRIPTION:
Test groups: 4 (400 subjects/group). 3 groups receiving 10-valent pneumococcal conjugate vaccine (3 different lots) as follows: - 10-valent vaccine (lot 1, 2 or 3) + DTPa combined vaccine; Control group receiving Prevenar + DTPa combined vaccine

ELIGIBILITY:
Inclusion criteria:

* Male or female between, and including, 6 and 12 weeks (42-90 days) of age at the time of the first vaccination, free of obvious health problems and with written informed consent obtained from the parent/guardian of the subject.

Exclusion criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceeding the first dose of study vaccine, or planned use during the study period.
* Planned administration/ administration of a licensed vaccine not foreseen by the study protocol during the period starting from one month before the first dose of vaccine(s) and during the entire study period.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1600
Dates: Start 2005-11; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Lot-to-lot consistency: antibody (Ab) concentrations to pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F and to carrier protein PD
Non-inferiority of 10-valent pneumococcal conjugate vaccine (pooled data of 3 10-Pn-PD-DiT vaccine groups) w.r.t. Prevenar: all anti-pneumococcal serotypes Ab concentrations>=0.20 µg/mL

SECONDARY OUTCOMES:
After each vaccination, occurrence of: solicited local, general symptoms within 4 days; | After each vaccination
Unsolicited adverse events within 31 days, SAEs (whole study period)
1m post dose3: For all vaccine pneumococcal serotypes: Opsono titres
Antibody (Ab) concentrations >= 0.20 µg/mL
Ab concentrations to protein D and seropositivity (S+) status
S+/seroprotection status to antigens in DTPa combo vaccine

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (34):
- Finland (14):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Jyväskylä
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Kotka
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vantaa
- France (14):
  - GSK Investigational Site, Bernay
  - GSK Investigational Site, Colombes
  - GSK Investigational Site, Courbevoie
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Dax
  - GSK Investigational Site, Draguignan
  - GSK Investigational Site, Essey-lès-Nancy
  - GSK Investigational Site, Le Havre
  - GSK Investigational Site, Maromme
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Nogent-sur-Marne
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Saint-Quentin
- Poland (6):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Trzebnica

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Chevallier B, Vesikari T, Brzostek J, Knuf M, Bermal N, Aristegui J, Borys D, Cleerbout J, Lommel P, Schuerman L. Safety and reactogenicity of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) when coadministered with routine childhood vaccines. Pediatr Infect Dis J. 2009 Apr;28(4 Suppl):S109-18. doi: 10.1097/INF.0b013e318199f62d. PMID 19325447
- [Background] Hausdorff WP, Dagan R, Beckers F, Schuerman L. Estimating the direct impact of new conjugate vaccines against invasive pneumococcal disease. Vaccine. 2009 Dec 9;27(52):7257-69. doi: 10.1016/j.vaccine.2009.09.111. Epub 2009 Oct 13. PMID 19833248
- [Background] Knuf M, Szenborn L, Moro M, Petit C, Bermal N, Bernard L, Dieussaert I, Schuerman L. Immunogenicity of routinely used childhood vaccines when coadministered with the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV). Pediatr Infect Dis J. 2009 Apr;28(4 Suppl):S97-S108. doi: 10.1097/INF.0b013e318199f61b. PMID 19325452
- [Background] Poolman J, Frasch C, Nurkka A, Kayhty H, Biemans R, Schuerman L. Impact of the conjugation method on the immunogenicity of Streptococcus pneumoniae serotype 19F polysaccharide in conjugate vaccines. Clin Vaccine Immunol. 2011 Feb;18(2):327-36. doi: 10.1128/CVI.00402-10. Epub 2010 Dec 1. PMID 21123523
- [Background] Schuerman L, Borys D, Hoet B, Forsgren A, Prymula R. Prevention of otitis media: now a reality? Vaccine. 2009 Sep 25;27(42):5748-54. doi: 10.1016/j.vaccine.2009.07.070. Epub 2009 Aug 8. PMID 19666154
- [Background] Schuerman L, Wysocki J, Tejedor JC, Knuf M, Kim KH, Poolman J. Prediction of pneumococcal conjugate vaccine effectiveness against invasive pneumococcal disease using opsonophagocytic activity and antibody concentrations determined by enzyme-linked immunosorbent assay with 22F adsorption. Clin Vaccine Immunol. 2011 Dec;18(12):2161-7. doi: 10.1128/CVI.05313-11. Epub 2011 Oct 12. PMID 21994351
- [Background] Vesikari T, Wysocki J, Chevallier B, Karvonen A, Czajka H, Arsene JP, Lommel P, Dieussaert I, Schuerman L. Immunogenicity of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) compared to the licensed 7vCRM vaccine. Pediatr Infect Dis J. 2009 Apr;28(4 Suppl):S66-76. doi: 10.1097/INF.0b013e318199f8ef. PMID 19325449
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 105553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 105553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 105553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 105553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 105553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 105553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register